CLINICAL TRIAL: NCT03100045
Title: A Phase I Study of Intra-Anally Administered Artesunate in Patients With High-Grade Anal Intraepithelial Neoplasia (AIN 2/3)
Brief Title: Intra-Anally Administered Artesunate in Patients With High-Grade Anal Intraepithelial Neoplasia (AIN 2/3)
Acronym: ART-AIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Frantz Viral Therapeutics, LLC (Industry); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090922
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: HPV-Related Anal Intraepithelial Neoplasia; AIN2/3; Artesunate; Alternative Treatment; Anal Dysplasia; Precancerous Conditions; Human Papilloma Virus
Keywords: HPV; suppository; Artesunate; artemisinin; anal dysplasia; treatment; alternative treatment; anal precancer; Johns Hopkins; Sandy Fang; Frantz Viral Therapeutics; Wisconsin; Evie Carchman
MeSH Terms: conditions — Precancerous Conditions | interventions — artemisinin

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled sequentially in each treatment cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ART 200 mg, 2 cycles (Experimental): Two five-day cycles of Artesunate suppositories, 200 mg/day
  Interventions: Drug: Artesunate Suppositories
- ART 200 mg, 3 cycles (Experimental): Three five-day cycles of Artesunate suppositories, 200 mg/day
  Interventions: Drug: Artesunate Suppositories
- ART 400 mg, 2 cycles (Experimental): Two five-day cycles of Artesunate suppositories, 400 mg/day
  Interventions: Drug: Artesunate Suppositories
- ART 400 mg, 3 cycles (Experimental): Three five-day cycles of Artesunate suppositories, 400 mg/day
  Interventions: Drug: Artesunate Suppositories
- ART 600 mg, 2 cycles (Experimental): Two five-day cycles of Artesunate suppositories, 600 mg/day
  Interventions: Drug: Artesunate Suppositories
- ART 600 mg, 3 cycles (Experimental): Three five-day cycles of Artesunate suppositories, 600 mg/day
  Interventions: Drug: Artesunate Suppositories

INTERVENTIONS:
Drug: Artesunate Suppositories — Artesunate suppositories for the treatment of (AIN2/3) Anal Intraepithelial Neoplasia
  Other Names: Artemisinin

SUMMARY:
This open label study investigates a novel non-surgical approach to the treatment of HPV-associated anal intraepithelial neoplasia, using Artesunate suppositories.

DETAILED DESCRIPTION:
Patients diagnosed with AIN 2/3 will be enrolled sequentially in treatment cohorts receiving different doses of Artesunate suppositories administered trans-anally. Doses of escalation will be 200 mg, 400 mg, and 600 mg. Treatment cohorts will consist of 2 or 3 cycles at each dose level. Suppositories will be administered daily for 5 days. Five days constitutes 1 cycle. Up to 3 cycles will be administered at Weeks 0, 2, and 4.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy-confirmed high-grade anal dysplasia (AIN 2, AIN 3, HSIL) by high resolution anoscopy (HRA)
* Female of childbearing potential: negative urine pregnancy test
* Able to provide informed consent
* Patients who have the ability to collaborate with planned follow-up (transportation, compliance history, etc.).
* Weight ≥50 kg.

Exclusion Criteria:

* Diagnosis of low-grade anal dysplasia (AIN 1, LSIL) by high resolution anoscopy
* Known anal, vulvar, cervical, or penile cancer
* CD4 count < 200 at the time of consideration for entry into this study
* Unable to provide informed consent
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.
* Patients who are on medical treatment with systemic immunosuppressants or steroids (e.g., active autoimmune disease)
* Extensive anal condyloma precludes the ability for the clinician to visualize HSIL during HRA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (Safety and tolerability) of Artesunate suppositories for the treatment of anal intraepithelial neoplasia (AIN2/3) | 6 weeks from the date of the first dosing
  Number of patients with serious adverse events or dose limiting toxicities related to the study medication, according to CTCAE4.0

SECONDARY OUTCOMES:
Number of patients with histologic regression of anal intraepithelial neoplasia (AIN2/3) to AIN1 or less | 16 weeks
  Number of patients with no AIN2/3 as assessed by high resolution anoscopy and biopsy
Number of patients with histologic regression of anal intraepithelial neoplasia (AIN2/3) to AIN1 or less | 28 weeks
  Number of patients with no AIN2/3 as assessed by high resolution anoscopy and biopsy
Number of patients with viral clearance of human papillomavirus (HPV) virus measured by HPV genotyping | 40 weeks
  Number of patients with HPV genotypes present at study entry which become undetectable during the study window

CONTACTS AND LOCATIONS:
Overall Officials: Sandy H Fang, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No